CLINICAL TRIAL: NCT05388851
Title: Education for Prevention of Melanoma in Hispanic Populations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-010065; NCI-2022-03769 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (Educational training) (Experimental): Participants complete an educational training module and complete questionnaire at baseline (before educational training module) and 3 months after completing educational training.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Complete educational training module
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This clinical trial is to develop an educational platform to educate and prevent melanoma in Hispanic populations. Melanoma is cancer arising in the skin. Educational platforms to increase the knowledge and practice of sun smart behaviors (sunscreen use, sun protective clothing use, self-skin examination) may help reduce risk of and incidence of melanoma and improve cancer survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop online education platform to educate the Hispanic community. II. Demonstrate improvement in knowledge and practice of sun smart behaviors. III. Determine if the education platform leads to increase visits to their medical provider and increase diagnosis of skin cancers, particularly melanoma, in our population.

OUTLINE:

Participants complete an educational training module and complete questionnaire at baseline (before educational training module) and 3 months after completing educational training.

ELIGIBILITY:
Inclusion Criteria:

* Mayo Clinic patients who self-identify as Hispanic or Latino
* Age 18 and older
* Have an email on file with Mayo Clinic

Exclusion Criteria:

* All patients who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Knowledge score after completing the educational module | Up to 3 months
  For quantitative variables, descriptive statistics including number of observations, mean, median, standard deviation, and range will be given for the values. Qualitative variables will be summarized using counts and percentages. Associations between quantitative variables will be conducted using the Pearson linear correlation coefficient, and the Chi-squared or Fisher's exact test for categorical variables.The melanoma knowledge score will be a percent correct, between 0% and 100% (100% is the best score), on a participant questionnaire. The primary outcome is the change in participant melanoma knowledge score before and immediately after completing the melanoma education (the intervention in this study).

SECONDARY OUTCOMES:
Knowledge score three months after completing the educational module | 3 months after completing education module
  For quantitative variables, descriptive statistics including number of observations, mean, median, standard deviation, and range will be given for the values. Qualitative variables will be summarized using counts and percentages. Associations between quantitative variables will be conducted using the Pearson linear correlation coefficient, and the Chi-squared or Fisher's exact test for categorical variables.The secondary outcome is their melanoma knowledge score at the three-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Mangold, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States